CLINICAL TRIAL: NCT06639867
Title: A Randomised Feasibility Study to Evaluate Home-based Personalised Virtual Reality Physiotherapy Rehabilitation Compared to Usual Care in the Treatment of Pain for People With Knee Osteoarthritis
Brief Title: Sensor-based Physiotherapy Intervention With Virtual Reality
Acronym: SPIN-VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Centre for Healthcare Evaluation, Device Assessment, and Research (CEDAR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPON1947-23
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Virtual reality; Physiotherapy; Home-based physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-based home physiotherapy (Experimental): Home-based non-immersive virtual reality using sensors strapped to the users limbs and body. They take part in a variety of games associated with movements of physiotherapy exercises.
  Interventions: Device: VR-based home physiotherapy
- Standard physiotherapy care (Active Comparator): Standard care as prescribed by the treating physiotherapist.
  Interventions: Other: Standard physiotherapy care

INTERVENTIONS:
Device: VR-based home physiotherapy — VR-based home physiotherapy
  Arms: VR-based home physiotherapy
Other: Standard physiotherapy care — Standard physiotherapy care as prescribed by the treating physiotherapist
  Arms: Standard physiotherapy care

SUMMARY:
This study is looking at the how the use of non-immersive virtual reality technology can be used to help people that have pain in their knees caused by osteoarthritis. It is a feasibility randomised controlled trial to investigate the feasibility of the use of the intervention by patients in their homes in a larger randomised controlled trial.

The intervention is a non-immersive virtual reality system. Through the use of painless sensors, patients are able to control an animated character on a screen through a series of games that replicates real physiotherapy exercises used to treat knee osteoarthritis. This intervention is being compared to a standard care physiotherapy programme.

As this is a feasibility study, it has no single primary outcome. Instead, the main outcome measures relate to feasibility of the study. This includes; feasibility of recruitment, completeness of outcome measures, the fidelity of healthcare professionals delivering the intervention, the acceptability of the intervention and trial procedures, adverse events, and adherence of the intervention.

Patients are randomised to receive either the intervention or control, and then spend 12-weeks in their assigned treatment. They then receive a 12-week and a 24-week follow up. Patient interviews are offered for those in the intervention arm to collect qualitative data regarding acceptability of the intervention and their participation in the study.

DETAILED DESCRIPTION:
This study is looking at the how the use of non-immersive virtual reality technology can be used to help people that have pain in their knees caused by osteoarthritis. It is a feasibility randomised controlled trial to investigate the feasibility of the use of the intervention by patients in their homes in a larger randomised controlled trial.

The intervention is a non-immersive virtual reality system. This involves sensors that are strapped to the user's arms, legs, head, or chest (depending on the specific exercise). Their movement then controls a character on the screen of either a laptop or a TV. Patients then work through a series of games that replicate physiotherapist exercises. Their performance in the games determines the difficulty of the games, and as patients improve, the exercises get harder. Patients are required to perform these exercises 3 times a week over 12 weeks. During this time, patients have the opportunity to attend clinics with a physiotherapist to review their progress. This intervention is being compared to standard care physiotherapy exercises that patients perform at home in their own time. This programme is prescribed to them by a physiotherapist, and they are followed up regularly over 12 weeks as they perform the programme at home.

This is a feasibility study, and has no single primary outcome or objective. Instead, there are several main outcomes and objectives related to the feasibility of the study and the intervention. The feasibility of recruitment to the study will be measured by the ability to achieve a recruitment of 4 patients per month, over 13 months. The recruitment target is 50. Patient willingness to be randomised will be measured by the reasons for non-consent and withdrawal given by patients. The completeness of outcome measures is measured by the of questionnaires and outcomes completed at 12- and 24-weeks post randomisation. The fidelity of healthcare professionals delivering the intervention will be measured by treatment logs for face-to-face contact, and the observation of two assessments for setting up knee osteoarthritis patients with the intervention. The acceptability of intervention and trial procedures to participants will be measured by interviews with patients and staff about expectations and experience of the intervention, and barriers and facilitators to trial participation. Adverse events experienced by participants from the intervention and trial procedures will also be measure by treatment logs. Adherence to the physiotherapy programme will be measured by the number of times and when patients logged in to the VR games and if follow up consultations were used. There are a variety of secondary objectives and outcome measures. A variety of measurements relating to muscle strength and endurance, aerobic capacity, exercise technique, central pain processing, and self-reported pain mechanisms and moderators will be used to understand how the exercises work to improve pain outcomes. The ability of the intervention to treat knee osteoarthritis will be measured by the OMERACT-OARSI core domain set, a variety of patient-reported outcome measures, pain sensitisation by algometer, and a dynamic balance using a step test.

The target population is adults with knee osteoarthritis who fulfil the NICE and ACR criteria for knee osteoarthritis diagnosis and who have been referred to a physiotherapy clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45 or older years
* Clinical diagnosis of knee osteoarthritis
* Referred for physiotherapy for clinically diagnosed knee osteoarthritis pain
* Activity related joint pain
* Self-reported knee pain on most days for the past 3 months
* Average pain severity in the past week of 4 or greater on a 10-point numeric rating scale
* Able to understand written and spoken English
* Able to provide written informed consent

Exclusion Criteria:

* Where knee is not identified by the participant as the main source of pain (e.g. comorbid painful conditions, widespread pain).
* Contraindication to exercise
* Pain caused by malignancy, fractures, or inflammatory arthritis
* Has received surgery for their knee pain in the last 12 months
* Has commenced another new treatment for knee pain, including intra-articular injection, during the preceding 12 weeks
* Concurrent ongoing treatment by physiotherapy other than the trial interventions
* Previous knee arthroplasty in either knee
* Unable to walk without a walking aid
* Unable or unwilling to engage in either active or control intervention

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 13-month recruitment period
  Ability to achieve a recruitment and randomisation of 4 patients per month, 50 patients within 13 months (number screened, consented, and randomised will be logged; reasons for non-consent or withdrawal will be recorded).
Completeness of outcome measures | 24-week follow up
  Number (%) of each questionnaire and mechanistic outcome completed at 12-weeks and 24-weeks post randomisation.
Fidelity of healthcare professionals delivering intervention | 12-week intervention period
  Treatment logs for face-to-face contact, observation of two assessments and training sessions for setting up patients with knee osteoarthritis with the intervention.
Acceptability of intervention and trial procedures | 12-week intervention period
  Interviews with patients and staff about expectations and experience of the intervention, and barriers and facilitators to trial participation.
Adverse events | 24-week follow up
  Treatment logs and patient interviews will be used to find issues related to knee symptoms or muscle soreness and falls, and motion sickness, plus any unexpected adverse events.
Adherence to the intervention | 12-week intervention period
  Number of times and date/time of when patients logged in to the VR games and number of physiotherapy follow-up consultations.

SECONDARY OUTCOMES:
Evaluate the processes for exercise mechanism of action at improving pain outcomes | 24-week follow up
  A variety of measurements relating to muscle strength and endurance, aerobic capacity, exercise technique, central pain processing, and self-reported pain outcomes and moderators.
Assess intervention to treat knee osteoarthritis | 24-week follow up
  The OMERACT-OARSI core domain set. A variety of patient-reported outcome measures. Pain sensitisation by algometer. Dynamic balance using a step test.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Cardiff University School of Healthcare Sciences, Cardiff
  - University Hospital of Wales, Cardiff

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Amri M, Bird S, Nistor DT, White J, Button K, Warner M, Walsh D, Shorten D, Evans R. Evaluating home-based personalised virtual reality physiotherapy rehabilitation compared with usual care in the treatment of pain for people with knee osteoarthritis: protocol for a randomised feasibility study. BMJ Open. 2025 Oct 21;15(10):e102994. doi: 10.1136/bmjopen-2025-102994. PMID 41125281